CLINICAL TRIAL: NCT03866876
Title: Umbilical Cord Arterial Eucapnic pH Compared With Arterial pH and Base Deficit as Predictor of Severe Adverse Outcomes Among Term Neonates
Brief Title: Eucapnic pH Compared With Arterial pH and Base Deficit
Acronym: PHE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: PHE
Record Dates: First submitted 2019-03-04; First posted 2019-03-07 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Neurologic Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hôpital Femme Mère Enfants births
  Interventions: Other: Eucapnic pH

INTERVENTIONS:
Other: Eucapnic pH — Collection of Biological marker (proposed by Racinet): eucapnic pH

SUMMARY:
Neonatal asphyxia per partum can be complicated by severe neurologic sequelae and can lead to neonatal death. Of the 0.2% of live births to cerebral palsy, 10 to 28% would be secondary to neonatal acidosis. Only metabolic acidosis plays a neurotoxic role, explaining the recent interest of Racinet et al. in the development of a new biochemical marker, more specific than pH or base deficit, of neonatal asphyxia per partum at risk of anoxo-ischemic encephalopathy. This eucapnic neonatal pH raises the hope of a biochemical marker of situations at risk of poor prognosis, with high diagnostic value, prognostic and forensic.

Our hypothesis is that eucapnic pH is more efficient than cord blood arterial pH and base deficit in the prediction of adverse neurologic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All birth more than 37 weeks of amenorrhea at the maternity ward of the hospital Femme-Mère-Enfant
* from 1st of january 2000 to 31 december 2016

Exclusion Criteria:

* Infants born out of the hospital and secondarily hospitalized in the hospital Femme-Mère-Enfant
* Children with congenital anomalies or without valid arterial and venous umbilical cord samples

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All birth more than 37 weeks of amenorrhea at the maternity ward of the hospital Femme-Mère-Enfant from 1st of january 2000 to 31 december 2016
Sampling Method: Non-Probability Sample
Enrollment: 36435 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients with at least one of these criteria including neonatal seizure, neonatal hypotonia requiring intensive care unit admission, neonatal encephalopathy, and/or neonatal death. | Between 2000 and 2016

CONTACTS AND LOCATIONS:
Overall Officials: Muriel DORET, Prof., Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Femme Mère Enfant, Bron, France